CLINICAL TRIAL: NCT03028441
Title: A Phase 1, Double Blinded, Placebo Controlled, Dose Comparison Trial to Evaluate the Safety, Immunogenicity and Schedule of Measles-Vectored Chikungunya Virus Vaccine (MV-CHIK) in Healthy Adults
Brief Title: Phase I Trial of Measles Vectored Chikungungya Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 15-0038; HHSN272201300015I
Record Dates: First submitted 2016-12-29; First posted 2017-01-23 (Estimated); Last update posted 2020-11-27 (Actual); Status verified 2017-10-12

CONDITIONS: Chikungunya Virus Infection
Keywords: Chikungunya; Immunogenicity; Measles; Vaccine
MeSH Terms: conditions — Chikungunya Fever; Measles

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Group 1- low dose (Experimental): 30 Subjects: 5 x 10^4 TCID50 MV-CHIK at Day1 and at Day 29 for 25 subjects, placebo for 5 subjects
  Interventions: Other: Placebo; Biological: VRC-CHKVLP059-00-VP
- Group 2-low dose (Experimental): 30 Subjects: 5 x 10^4 TCID50 MV-CHIK at Day 1 and at Day 85 for 25 subjects, placebo for 5 subjects
  Interventions: Other: Placebo; Biological: VRC-CHKVLP059-00-VP
- Group 3-low dose (Experimental): 30 Subjects: 5 x 10^4 TCID50 MV-CHIK at Day 1and at Day 169 for 25 subjects, placebo for 5 subjects
  Interventions: Other: Placebo; Biological: VRC-CHKVLP059-00-VP
- Group 4 -high dose (Experimental): 30 Subjects: 5 x 10^5 TCID50 MV-CHIK at Day 1 and at Day 29 for 25 subjects, placebo for 5 subjects
  Interventions: Other: Placebo; Biological: VRC-CHKVLP059-00-VP
- Group 5-high dose (Experimental): 30 Subjects: 5 x 10^5 TCID50 MV-CHIK at Day 1and at Day 85 for 25 subjects, placebo for 5 subjects
  Interventions: Other: Placebo; Biological: VRC-CHKVLP059-00-VP
- Group 6-dose-High Dose (Experimental): 30 Subjects: 5 x 10^5 TCID50 MV-CHIK at Day 1and at Day 169 for 25 subjects, placebo for 5 subjects
  Interventions: Other: Placebo; Biological: VRC-CHKVLP059-00-VP

INTERVENTIONS:
Other: Placebo — Placebo
Biological: VRC-CHKVLP059-00-VP — Measles-vectored Chikungunya vaccine

SUMMARY:
This study is a randomized, double-blinded, Phase 1, placebo- controlled, and dose comparison trial to evaluate the safety, immunogenicity and schedule of MV-CHIK. Two dosage levels and 3 immunization schedules will be evaluated. This study will enroll up to 180 healthy subjects aged 18 to 45 years.Study duration is approximately 22 months. Subject participation duration is approximately 8-13 months. The primary objectives are to evaluate the safety and tolerability of 5 x 10^4 TCID50 and 5 x 10^5 TCID50 MV-CHIK and placebo following two consecutive intramuscular injections and to assess the CHIKV serum plaque reduction neutralization test (PRNT50) antibody responses to 5 x 10^4 TCID50, 5 x 10^5 TCID50 of MV-CHIK or placebo on day 29 following the first dose.

DETAILED DESCRIPTION:
This study is a randomized, double-blinded, Phase 1, placebo- controlled, and dose comparison trial to evaluate the safety, immunogenicity and schedule of MV-CHIK. Two dosage levels (5 x 10^4 or 5 x 10^5 TCID50) and 3 immunization schedules (days 1 and 29, days 1 and 85 or days 1 and 169) will be evaluated. The study will have 6 cohorts, each with 30 subjects, 25 of whom will receive study vaccine and 5 of whom will receive placebo. Cohorts 1-3 will receive the low dosage of the lyophilized vaccine product (5 x 10^4 TCID50) and cohorts 4-6 will receive the high dosage (5 x 10^5 TCID50) of the lyophilized vaccine product. Each subject will receive two study injections using one of the three dosing schedules outlined above. This study will enroll up to 180 healthy subjects aged 18 to 45 years (inclusive). Subjects will be counseled on the study and will then sign an informed consent prior to any study procedures. Screening will be performed which will include evaluation of medical history, travel history to countries with known CHIKV circulation, medication history, a physical examination and safety laboratory evaluations. Study duration is approximately 22 months. Subject participation duration is approximately 8-13 months. The primary objectives are to evaluate the safety and tolerability of 5 x 10^4 TCID50 and 5 x 10^5 TCID50 MV-CHIK and placebo following two consecutive intramuscular injections and to assess the CHIKV serum plaque reduction neutralization test (PRNT50) antibody responses to 5 x 10^4 TCID50, 5 x 10^5 TCID50 of MV-CHIK or placebo on day 29 following the first dose. The secondary objectives are to assess the CHIKV serum plaque reduction neutralization test (PRNT50) antibody responses to 5 x 10^4 TCID50, 5 x 10^5 TCID50 MV-CHIK and or placebo using three dose schedules (days 1 and 29, days 1 and 85, or days 1 and 169) on day 29 following the second dose, assess CHIKV serum PRNT50 antibody responses to 5 x 10^4 TCID50, 5 x 10^5 TCID50 MV-CHIK or placebo on days 15, 85 and 169 following the second dose of vaccine, assess the CHIKV serum ELISA antibody responses to 5 x 10^4 TCID50, 5 x 10^5 TCID50 MV-CHIK or placebo on day 29 following the first dose of vaccine and days 15, 29, 85 and 169 following the second dose of vaccine, and to assess the durability of CHIKV serum ELISA and PRNT50 antibody responses to 5 x 10^4 TCID50, 5 x 10^5 TCID50 MV-CHIK or placebo on day 85 (Groups 2+5) and day 169 (Groups 3+6) following the first dose of vaccine.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria must be assessed by a clinician licensed to make medical diagnoses. Subjects must meet all of the following inclusion criteria to participate in this study

1. Males and non-pregnant females between the ages of 18 and 45 years (at study start), inclusive.
2. Provide written informed consent before initiation of any study procedures.
3. Women of childbearing potential must agree to practice adequate contraception during the 30 days prior to Day 1, the first injection, through 85 days after the second study injection. A woman is considered of childbearing potential unless surgically sterile (tubal ligation, bilateral oophorectomy, or hysterectomy) or post-menopausal (> /= 1 year) or successful Essure placement (permanent, non-surgical, non-hormonal sterilization) with documented confirmation test at least 3 months after the procedure. Acceptable birth control methods include but are not limited to: abstinence from sexual intercourse with men; monogamous relationship with a vasectomized partner; double-barrier methods (condoms, diaphragms, spermicides; and intrauterine devices); and licensed hormonal methods.
4. In good health, as judged by the investigator and determined by vital signs, medical history, and a physical examination. Temperature 37.8°C, heart rate 50-110bpm (inclusive), systolic blood pressure 85-150 mmHg (inclusive), diastolic blood pressure 55-95 mmHg (inclusive). Subjects may be on chronic or as needed (prn) medications if, in the opinion of the site principal investigator or appropriate sub-investigator, they pose no additional risk to subject safety or assessment of reactogenicity and immunogenicity. NOTE: Athletically trained subjects with a pulse > \= 45 - 49 may be enrolled if an ECG shows no evidence of first, second or third degree heart block.
5. Screening laboratory values must be within site normal limits, though trace urine protein is acceptable. Screening labs will include: Blood hemoglobin, White blood cell (WBC) count, Absolute neutrophil count, Platelets, Creatinine, Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), Bilirubin (total), Glucose (random, must be less than 140), Urine dipstick for protein and glucose (negative to trace protein are acceptable), Negative HIV 1/2 antibody/antigen test, Hepatitis B surface antigen (HBsAg), and Hepatitis C virus (HCV) antibody NOTE: Creatinine values lower than the normal range may be acceptable if the PI or a designated licensed clinician determines that these laboratory findings are not clinically significant. HIV and hepatitis C viral load PCR testing may be performed for individuals suspected of having indeterminate antibody/antigen testing (Sites will use the standard HIV testing protocol for their institution).
6. Able to understand and comply with planned study procedures and willing to be available for all study-required procedures, visits and calls for the duration of the study.
7. Willing to abstain from donating whole blood or blood derivatives until 90 days after the final study injection.
8. History of measles vaccination.

Exclusion Criteria:

1. History of known chikungunya infection.
2. Previous vaccination with an investigational chikungunya vaccine.
3. Past residence in, or travel for greater than 1 consecutive month within the past 6 months to, a location known to have local CHIKV transmission. (Examples of countries with local chikungunya virus transmission include, but are not limited to, countries in sub-Saharan Africa, South Asia, the Indian and Pacific Ocean). Residence in or travel to Central and South America, the Caribbean, Florida, Puerto Rico and the U.S. Virgin islands, if prior to 2013, will be permitted.
4. Plan to travel to a location known to have local CHIKV transmission during the course of the study or history of travel to one of these countries within 30 days prior to screening. Travel to Florida will be permitted. Those planning travel to Florida will be provided information on mosquito bite protection.
5. Body temperature >/ =100 °F (>/ =37.8°C) or acute illness within 3 days before study injection days (subject may be rescheduled).
6. A positive serum or urine pregnancy test at screening or within 24 hours prior to study injection, women who are planning to become pregnant, or women who are breastfeeding. If female of childbearing potential as defined in Inclusion Criterion 3. From 30 days prior to entering the study until 85 days after the final study injection.
7. Any clinically significant acute or chronic medical condition that, in the opinion of the investigator, would preclude participation. E.g., History of seizure disorders (other than febrile seizures as an infant), autoimmune disease, immunodeficiency, any spleen disease, active malignancy, active asthma, known cardiac disease, pulmonary disease, liver disease, renal disease, unstable or progressive neurological disorders, diabetes mellitus, and transplant recipients.
8. History of thrombocytopenia, idiopathic thrombocytopenic purpura or other platelet disorder.
9. A history of chronic arthritis or chronic arthralgia symptoms.
10. Used an immunosuppressive or immunomodulatory drug for 2 or more consecutive weeks within 6 months prior to the first study injection (nasal and topical steroids are allowed). Such as >/ =20 mg total dose/day of prednisone orally or > 840 µg of inhaled beclomethasone.
11. A diagnosis of schizophrenia, bipolar disease, or history of hospitalization for a psychiatric condition or previous suicide attempt.
12. A history of treatment for any other psychiatric disorder in the past 3 years that increases the risk to the subject in the opinion of the investigator Treatment for mild depression or anxiety using a single antidepressant or anti-anxiety medication will be allowed so long as the subject has been on stable doses for 3 months.
13. Received immunoglobulin or other blood product within 3 months prior to enrollment or planned receipt of immunoglobulin or a blood product through study day 169 following the second dose of vaccine.
14. Received or plan to receive any live licensed vaccines within 4 weeks or inactivated licensed vaccines within 2 weeks of any study injection.
15. Received or plans to receive measles-containing vaccine within 3 months prior to enrollment or planned to receive through study day 29 following the second dose of vaccine. measles, mumps, rubella vaccine.
16. History of anaphylaxis or severe allergic reaction to vaccines or history of allergic reaction to any components in the MV-CHIK vaccine.
17. Received an experimental or investigational agent within 1 month before study injections or expectation to receive an experimental agent through 6 months following the last study injection. Vaccine, drug, biologic, device, blood product, or medication.
18. Any condition that would, in the opinion of the investigator, place the subject at an unacceptable injury risk, render him/her unable to meet the requirements of the protocol, or that may interfere with successful study completion.
19. A history of alcohol or drug abuse during the previous 3 years For example, daily excessive alcohol or marijuana use or frequent binge drinking as determined by the investigator.
20. Presence of tattoos that, in the opinion of the investigator, would preclude evaluation of the injection site.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2019-01-17 (Actual)

PRIMARY OUTCOMES:
CHIKV serum antibody Geometric Mean Titer using PRNT50 | On Day 29 post dose 1
Mean fold change in PRNT50 anti-CHIKV antibody responses | On Day 29 post dose 1
The number of solicited injection site reactions | Day 1 through Day 15 following both study injections
The number of solicited systemic reactions | Day 1 through Day 15 following both study injections
The number of vaccine-related serious adverse events | Day 1-660
The number of vaccine-related unsolicited adverse events | Day 1 through Day 29 following each study vaccination
The proportion of subjects with at least a 4-fold increase in CHIKV serum antibody titer, using PRNT50 (Plaque Reduction Neutralization Test) | On Day 29 post dose 1

SECONDARY OUTCOMES:
anti-CHIKV antibody Geometric Mean Titer using ELISA and PRNT anti-CHIKV antibody responses levels (groups 2 and 5 | On Day 85
Anti-CHIKV antibody Geometric Mean Titer using in ELISA and PRNT anti-CHIKV antibody responses levels (groups 3 and 6) | On Day 169
CHIKV serum antibody Geometric Mean Titer using ELISA | On Day 29 following the first dose
CHIKV serum ELISA antibody Geometric Mean Titer | On Day 15, 29, 85, and 169 following the second dose
CHIKV serum PRNT50 antibody Geometric Mean Titer | On Day 15, 85, and 169 following the second dose
CHIKV serum PRNT50 antibody Geometric Mean Titer | On Day 29 following the second dose
Mean fold change from baseline to CHIKV using ELISA and PRNT anti-CHIKV antibody responses levels (groups 2 and 5) | On Day 85
Mean fold change from baseline to CHIKV using in ELISA and PRNT anti-CHIKV antibody responses levels (groups 3 and 6) | On Day 169
Mean fold change to CHIKV in ELISA anti-CHIKV antibody responses | On Day 15, 29, 85, and 169 following the second dose
Mean fold change to CHIKV in ELISA anti-CHIKV antibody responses | On Day 29 following the first dose
Mean fold change to CHIKV in PRNT50 anti-CHIKV antibody responses | On Day 15, 85, and 169 following the second dose
Mean fold change to CHIKV in PRNT50 anti-CHIKV antibody responses | On Day 29 following the second dose
The proportion of subjects with at least a 4-fold increase in anti-CHIKV antibody titer using ELISA and PRNT anti-CHIKV antibody responses levels (groups 2 and 5) | On Day 85
The proportion of subjects with at least a 4-fold increase in anti-CHIKV antibody titer using ELISA and PRNT anti-CHIKV antibody responses levels (groups 3 and 6) | On Day 169
The proportion of subjects with at least a 4-fold increase in CHIKV serum antibody titer, using ELISA | On Day 29 following the first dose
The proportion of subjects with at least a 4-fold increase in CHIKV serum ELISA antibody titer | On Day 15, 29, 85, and 169 following the second dose
The proportion of subjects with at least a 4-fold increase in CHIKV serum PRNT50 antibody titer | On Day 15, 85, and 169 following the second dose
The proportion of subjects with at least a 4-fold increase in CHIKV serum PRNT50 antibody titer | On Day 29 following the second dose

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Emory Children's Center - Pediatric Infectious Diseases, Atlanta, Georgia
  - University of Iowa - Vaccine Research and Education Unit, Iowa City, Iowa
  - Baylor College of Medicine - Molecular Virology and Microbiology, Houston, Texas